CLINICAL TRIAL: NCT06241027
Title: Effects of Myofascial Release and Nerve Flossing Technique on Pain and Disability in Patients With Lumbar Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0234
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Lumbar Radiculopathy
Keywords: Lumbar radiculopathy, Myofascial release, Nerve flossing
MeSH Terms: conditions — Radiculopathy | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nerve flossing technique (Experimental): Nerve flossing technique will be repeated 3 times a week for 15 minutes per session include 2 sets of 10 repetitions for 4 weeks
  Interventions: Other: Nerve flossing technique
- Myofascial release (Experimental): Myofascial release technique will be given to the patients 3 times a week for 10 minutes with a total 4 weeks of treatment plan.
  Interventions: Other: Myofascial release

INTERVENTIONS:
Other: Nerve flossing technique — The nerve flossing technique will be perform actively with the participant sitting on the chair. The participant flexed the knee of the target lower extremity backward beside the chair as far back as possible and flexed the neck at the same time, holding both the flexed knee and neck in thisposition for 5 seconds. The participant in turn extended the neck and knee of the target lower extremity, abducted and flexed the hip until pain will feel and did not push beyond that point. This extended position will be hold for 5 seconds.
  Arms: Nerve flossing technique
Other: Myofascial release — Myofascial release therapy involved the application of a low load, long duration stretch along the line of maximal fascial restriction. Pressure will be applied directly on the skin toward the direction of restriction until resistance of the tissue barrier will felt, Once found , the collagenous barrier will engaged for 90-120 seconds without sliding over the skin or forcing the tissues until the fascia complex started to yield and a sensation of softening will achieved.This stage will be repeated up to 5 times for new barrier until the sensation of tissue restriction during stretching became weaker.
  Arms: Myofascial release

SUMMARY:
Radiculopathy is a clinical condition which involves one or more nerves resulting in impaired function. The site of injury in radiculopathy is at the level of the spinal nerve root. The result is pain known as radicular pain, weakness in limb, numbness, paresthesia and difficulty in controlling specific muscles. The objective of the study will be to see the effects of myofacsial release and nerve flossing technique on pain and disability in patients with lumbar radiculopathy.

DETAILED DESCRIPTION:
This study will be randomized controlled trail. Participants having age in between 20-45 with low back pain radiating to the lower leg from last 2 months will be included in the study while the participants with lumbar spinal fracture, lumbar spinal tumor, peripheral vascular disease and systemic disease will be excluded from the study. Total 36 number of participants will be included in the study by non probability convenient sampling that will be randomly allocated into two groups by lottery method. Group A will receive nerve flossing technique and myofascial release along with conventional treatment while group B will receive nerve flossing technique along with conventional treatment. Nerve flossing technique will be given to patients 3 times per week for 15 minutes per session. Myofascial release technique will be given to the patients 3 times a week for 10 minutes with a total 4 weeks of treatment plan. All the participants will undergo a pre and post treatment test via numeric pain rating scale which will be used for rating pain, SLR, oswestry disability index which will be used for rating the level of disability. The importance of the study is to investigate the effects of these techniques in a controlled research setting will help determine their potential role in personalized treatment plans for patients with lumbar radiculopathy. The data will be analyzed via SPSS version 23.

ELIGIBILITY:
Inclusion Criteria: The age of patients in between 20-45 years old, Patients with low back pain radiating to the lower leg from the last 2 month, patients with positive straight leg raise test.

-

Exclusion Criteria: Patients with lumbar spinal fracture, patients having spinal tumor, patients with unhealed wound on the lumbosacral area, patients having peripheral vascular disease, patients who diagnosed with systemic disease such as diabetes mellitus and rheumatoid arthritis.

-

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-02-12 (Estimated); Study Completion 2024-02-12 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale | 4 weeks
  This scale rates the level of pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme.

SECONDARY OUTCOMES:
Straight leg raise test | 4 weeks
  The Straight Leg Raise (SLR) test is to identify disc pathology or nerve root irritation, as it mechanically stresses lumbosacral nerve roots.

OTHER OUTCOMES:
Oswestry disability index questionnaire | 4 weeks
  This questionnaire provides information as to how your back pain has affected your ability to manage everyday life and check the level of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Asrar Yousaf, Phd, Principal Investigator — Riphah International University
Locations (1):
- Ripha international university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No